CLINICAL TRIAL: NCT07310667
Title: Assessing the Relationship Between Frailty and Skeletal Muscle Thickness in Critically Ill Patients: A Prospective Observational Study.
Brief Title: Assessing the Relationship Between Frailty and Skeletal Muscle Thickness in Critically Ill Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayşe EKEN, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: 13.03.2025_E25-423
Record Dates: First submitted 2025-06-25; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Fraility; Nutrition Assessment; Ultrasound Evaluation; Critical Illness
Keywords: Fraility; Nutrition Assessment; Muscle Ultrasound; Muscle Thickness; Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Muscle ultrasound — Examine all patients both USG and Fraility scale
  Other Names: Fraility Scale

SUMMARY:
Assessment of muscle mass in critically ill patients is critical for both improving clinical outcomes and monitoring the effectiveness of nutritional interventions. Loss of muscle mass is associated with mortality and morbidity in the elderly, including organ transplantation, trauma, and sepsis. Previous studies have assessed muscle mass using computed tomography. The use of computed tomography is costly, carries radiation risks, and requires the patient to be transported to a CT scanner. In contrast, ultrasonography is a noninvasive, rapid, and bedside method without radiation exposure. In particular, anterior thigh muscle thickness (ATMT) stands out as a reliable biomarker in the assessment of muscle mass. ATMT measurement includes the assessment of the combined depth of the vastus intermedius and rectus femoris muscles in the anterior thigh. There is no study in the literature examining the effects of anterior thigh muscle thickness measured by ultrasonography on malnutrition and frailty in intensive care patients. In this study, we aimed to investigate the effects of anterior thigh muscle thickness on frailty, malnutrition and length of stay in intensive care patients.

DETAILED DESCRIPTION:
According to the World Health Organization, the global elderly population is rapidly increasing, and this is causing a significant increase in the number of elderly patients admitted to intensive care units (ICUs). The rate of individuals aged 60 and over, which was 12% in 2015, is estimated to reach 22% in 2050. This demographic change significantly increases the use of intensive care beds and the duration of healthcare services by frail and vulnerable elderly individuals. Malnutrition, frailty and mortality rates in patients hospitalized in intensive care units are among the main factors that directly affect patient prognosis. Malnutrition negatively affects both short- and long-term clinical outcomes by causing serious consequences such as weakening of the immune system, increased susceptibility to infections, delayed wound healing and decreased muscle mass. Frailty is characterized by the decrease in physiological reserves due to age and disease and has an important role in predicting clinical deterioration in intensive care patients.

The aim of our study was to investigate the effects of anterior thigh muscle thickness on frailty, malnutrition, and length of stay in intensive care in intensive care patients.

This study was designed as a prospective, observational study. The study will be conducted on patients admitted to the Ankara Education and Research Hospital Anesthesia intensive care unit for any reason after obtaining ethics committee approval.

ELIGIBILITY:
Inclusion Criteria:

* over 65
* 1 week min stay

Exclusion Criteria:

* Patients under 65 years of age
* those with cardiac arrest, terminal illnesses, advanced cancer, advanced neurodegenerative diseases,
* those with knee or hip prosthesis that would affect the anterior thigh muscle thickness measurement those whose intensive care stay did not exceed 1 week will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Over 65 years, critically ill patients, who are submitted to ICU.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Front Thigh Muscle Measurement | Ultrasound assessments will be performed within 24 hours of intensive care unit (ICU) admission and repeated on ICU days 3 and 7.
  Anterior thigh muscle thickness will be measured using ultrasonography with a linear transducer operating at 5-10 MHz. Using ample gel and minimal probe compression, the measurement site will be marked at the midpoint between the anterior superior iliac spine (SIAS) and the superior pole of the patella. Total quadriceps thickness-defined as the combined thickness of the rectus femoris and vastus intermedius-will then be recorded. Thickness will be measured as milimeter. Ultrasound assessments will be performed within 24 hours of intensive care unit (ICU) admission and repeated on ICU days 3 and 7.
Frailty Assessment | Frailty will be ascertained at ICU admission by interviewing family/caregivers about the patient's frailty level prior to the acute illness and hospitalization.
  Frailty will be assessed using the Clinical Frailty Scale (CFS). Frailty status will be determined at the time of ICU admission by interviewing family members/caregivers to ascertain the patient's frailty level prior to the acute illness and hospitalization.
  Clinical Frailty Scale (CFS):
  1 Very fit; 2 Well; 3 Managing well; 4 Vulnerable-independent but slowed, fatigued; 5 Mildly frail-needs help with instrumental ADLs (finances, transport, heavy housework, meds); 6 Moderately frail-needs help with all outside activities/housework; may need minimal help bathing/dressing; 7 Severely frail-dependent for personal care but clinically stable; 8 Very severely frail-dependent, near end of life; 9 Terminally ill-life expectancy <6 months. Classification: 1-3 non-frail; 4 pre-frail; ≥5 frail
Nutritional Status Assessment | Will be ascertained at ICU admission by interviewing with family/caregivers
  Assessment nutritional risk in ICU patients and identify those at high risk of malnutrition, the NRS-2002, GLIM criteria, and the NUTRIC score will be used.
  (NRS-2002: Nutritional Risk Screening 2002; GLIM: Global Leadership Initiative on Malnutrition; NUTRIC: Nutrition Risk in the Critically Ill.)

SECONDARY OUTCOMES:
Critical Care Scoring System: APACHE II | During the first 24 hours of ICU admission
  The APACHE II (Acute Physiology and Chronic Health Evaluation II) score is a system used to assess mortality risk in ICU patients. It will be calculated from physiologic and clinical parameters obtained during the first 24 hours of ICU admission. The score is based on acute physiologic variables, age, and chronic health status, and ranges from 0 to 71.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training And Research Hospital, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: between January 1st 2026 and May 1st 2026

REFERENCES:
- [Background] Bruno RR, Wernly B, Bagshaw SM, van den Boogaard M, Darvall JN, De Geer L, de Gopegui Miguelena PR, Heyland DK, Hewitt D, Hope AA, Langlais E, Le Maguet P, Montgomery CL, Papageorgiou D, Seguin P, Geense WW, Silva-Obregon JA, Wolff G, Polzin A, Dannenberg L, Kelm M, Flaatten H, Beil M, Franz M, Sviri S, Leaver S, Guidet B, Boumendil A, Jung C. The Clinical Frailty Scale for mortality prediction of old acutely admitted intensive care patients: a meta-analysis of individual patient-level data. Ann Intensive Care. 2023 May 3;13(1):37. doi: 10.1186/s13613-023-01132-x. PMID 37133796
- [Background] Lee ZY, Ong SP, Ng CC, Yap CSL, Engkasan JP, Barakatun-Nisak MY, Heyland DK, Hasan MS. Association between ultrasound quadriceps muscle status with premorbid functional status and 60-day mortality in mechanically ventilated critically ill patient: A single-center prospective observational study. Clin Nutr. 2021 Mar;40(3):1338-1347. doi: 10.1016/j.clnu.2020.08.022. Epub 2020 Aug 28. PMID 32919818
- [Background] Kalaiselvan MS, Yadav A, Kaur R, Menon A, Wasnik S. Prevalence of Frailty in ICU and its Impact on Patients' Outcomes. Indian J Crit Care Med. 2023 May;27(5):335-341. doi: 10.5005/jp-journals-10071-24456. PMID 37214110